CLINICAL TRIAL: NCT03942874
Title: Development and Initial Tests of Reward Re-Training: A Novel Treatment For Reward Dysfunction
Acronym: Recharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Adrienne Juarascio, Assistant Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project Recharge
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Binge Eating; Binge-Eating Disorder; Bulimia Nervosa
Keywords: reward; reward dysfunction; group treatment; binge eating
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will complete baseline sessions and then complete treatment right away.
  Interventions: Behavioral: Group Reward Retraining
- Waitlist Control (Experimental): Participants will complete a baseline session and then wait for 10 weeks before starting treatment.
  Interventions: Behavioral: Group Reward Retraining

INTERVENTIONS:
Behavioral: Group Reward Retraining — Adapted behavioral activation group treatment for binge eating with values and cognitive skills integrated
  Other Names: behavioral activation

SUMMARY:
The purpose of this study is to test a novel treatment for binge eating that will be compared to a waitlist control group. The investigators are seeking to target factors that might influence binge eating by increasing reward in non-food life domains. The treatment is weekly for 10 weeks and will take place at Drexel University in Philadelphia.

DETAILED DESCRIPTION:
At the start of the study, you will be interviewed to determine if you are eligible to participate in the study.

Once you are determined to be eligible, you will be assigned at random to a treatment group or a waitlist control group. The chances of being assigned to each condition are like a flip of a coin. If you are placed in the waitlist control group, you will complete a 10-week waiting period after your initial assessment, then complete another assessment and treatment after 10 weeks.

First, the study will be explained to you and you will be given an opportunity to ask questions about the study and sign this consent form.

You will complete the baseline assessment, which will take place in 2 sessions. The first session will take place at Drexel and will include behavioral tasks and surveys. The second session will take place at Temple University and will include an fMRI (functional magnetic resonance imaging) scan. Both sessions combined will take about 6 hours total. This baseline assessment will involve: Behavioral tasks: These are designed to measure your responses to food reward and other pleasant events. These tasks will be in the form of computer games where you will rate and sort different rewarding items. These will take place at Drexel University. Surveys: questions regarding demographics, disordered eating, weight history, and other psychological symptoms. These will take place at home if you choose to complete them before your assessment, or at Drexel University. fMRI task: fMRI scans will take place at Temple University. After consenting, an fMRI technician will review the safety checklist to make sure you have no metal objects in your clothing or on your body that might enter the scanner. Following this review, you will be taken to the MRI scanner. The scan will take about 1-hour. You will be asked to lie on your back on the scanner bed. You will be fit with a set of headphones, a microphone and goggles that are connected to a computer display. You will have continuous contact with the research team using the headphone and microphone. At any time during scanning, you can ask to be taken out of the scanner. The study involves lying quietly in the scanner, viewing pictures and hearing sounds while selecting answers to questions presented on the computer display. The scanning will also include a structural scan. If the computer procedures work well, the entire scanning session should last no longer than 60 minutes. Even if the scanning is not complete, you will be taken out of the scanner after 60 minutes.

You can expect to interact in group therapy with other study participants, led by Drexel faculty and graduate students in private rooms at the Psychology Department of Drexel University. You will receive 10 sessions of weekly group treatment that are each approximately one hour in length. You will complete the same assessment procedure you completed at the beginning of treatment at mid-treatment (after session 5-with the exception of the fMRI tasks) and post-treatment (after session 10). All sessions and assessments will be audio-recorded and securely stored until the completion of study analyses. If you do not wish to be audio-recorded, you may not participate in the study. If you are withdrawn from the study and wish for your recordings to be deleted, you may request that the researchers delete them.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant binge eating

Exclusion Criteria:

* non-removable metal object in body
* non-removable hair extensions or wig
* tattoo above shoulders
* significant amounts of metal fillings in mouth
* BMI below 18.5
* BMI above 40
* Currently experiencing severe psychopathology that would limit their ability to engage in study (e.g. suicidality, substance use disorder, psychotic disorder)
* Are unable to fluently speak, write and read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Feedback Questionnaire (FQ) | Assessed at mid- and post- treatment sessions (3 months)
  The feedback questionnaire asks qualitative questions about the quality of and satisfaction with the treatment. The feedback questionnaire does not report either subscale scores or a total score. The FQ will be used to obtain qualitative acceptability ratings.
Binge frequency assessed by the Eating Disorder Examination | Change from baseline assessment (before beginning treatment) to post-treatment assessment (10 weeks after baseline assessment)
  Frequency (number of days and number of instances) of binge eating behaviors over the past 28 days assessed by the Eating Disorder Examination

SECONDARY OUTCOMES:
Reward responsivity to natural (nonfood) reward- Reward Probability Index (RPI) | Change from baseline assessment (before beginning treatment) to post-treatment assessment (10 weeks after baseline assessment)
  The Reward Probability Index is a 20-item self-report measure of reward. The measure yields a total score. The total score is computed by summing responses, so the possible score range is 20 to 80. For the total score, higher scores indicate greater reward. The RPI will be used to assess increase in responsivity to nonfood reward.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Juarascio, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel WELL Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juarascio AS, Presseller EK, Wilkinson ML, Kelkar A, Srivastava P, Chen JY, Dengler J, Manasse SM, Medaglia J. Correcting the reward imbalance in binge eating: A pilot randomized trial of reward re-training treatment. Appetite. 2022 Sep 1;176:106103. doi: 10.1016/j.appet.2022.106103. Epub 2022 Jun 1. PMID 35662619